CLINICAL TRIAL: NCT07051460
Title: MULTISENSORIALIDAD Y BOCA Estudio Del Efecto de estímulos Propioceptivos en el área estomatognática Sobre la percepción Visual, Con y Sin Sonido
Brief Title: Study of the Effect of Proprioceptive Stimuli in the Stomatognathic Area on Visual Perception, With and Without Sound
Status: Completed | Type: Observational
Sponsor: Sophie Román Richon (Other)
Collaborators: Hospital Odontològic UB (Other)
Responsible Party: Sponsor-Investigator, Sophie Román Richon, Associate Professor Department of Odontostomatology, University of Barcelona
Organization: University of Barcelona (Other)
Other Study IDs: CEIm HOUB 43/2022
Record Dates: First submitted 2025-06-12; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Proprioception; Visual Perception; Multisensory; Stomatognathic System
Keywords: Proprioception; Multisensory Integration; Trigeminal Nerve; Visual Perception; Periodontal Mechanoreceptors; Stomatognathic System
MeSH Terms: interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic; Clinical Trials, Phase III as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy young adult participants (ages 20-29) underwent a 4-phase experimental protocol involving auditory and oral proprioceptive stimuli under controlled conditions, using the Vertical Maddox Test to assess transient visual changes.
  Interventions: Other: Baseline Condition (No Stimuli); Other: Auditory Stimulation only; Other: Auditory and Oral Proprioceptive Stimulation (OPS); Other: Oral Proprioceptive Stimulation Only (OPS)

INTERVENTIONS:
Other: Baseline Condition (No Stimuli) — Participants underwent baseline evaluation using the Vertical Maddox Test with no auditory or oral proprioceptive stimulation. This phase was used to confirm the absence of spontaneous visual pseudo-scotomas and served as an internal control condition for each participant.
  Other Names: Phase 1
Other: Auditory Stimulation only — Participants received bilateral auditory stimulation consisting of 500 Hz tones (500 ms duration, 50 dB) delivered through wireless headphones, without any accompanying oral stimuli. This condition was used to assess the isolated effect of sound on visual perception using the Vertical Maddox Test.
  Other Names: Phase 2
Other: Auditory and Oral Proprioceptive Stimulation (OPS) — Participants received simultaneous auditory and oral proprioceptive stimuli while undergoing the Vertical Maddox Test. - Auditory: 500 Hz tones (500 ms, 50 dB) via headphones. - Oral Proprioceptive Stimuli (OPS): included Combined Oral Stimuli (e.g., tongue and lip self-administered positions) and Dental Stimuli (mechanical pressure or traction on central incisors using a calibrated probe). This condition aimed to assess whether OPS could modulate or eliminate sound-induced visual pseudo-scotomas.
  Other Names: Phase 3
Other: Oral Proprioceptive Stimulation Only (OPS) — Participants received oral proprioceptive stimuli alone, without auditory input, during the Vertical Maddox Test. - Combined Oral Stimuli (COS): self-administered tongue/lip positions. - Dental Stimuli (DS): applied by the operator to central incisors. This condition was used to evaluate the independent effect of OPS on visual perception.

SUMMARY:
The goal of this observational study is to investigate how oral proprioceptive stimuli affect visual perception and auditory-visual integration in healthy young adults. The main questions it aims to answer are:

* Can Oral Proprioceptive Stimuli (OPS) induce Visual pseudo-Scotomas (VS) in the absence of other stimuli?
* Can Oral Proprioceptive Stimuli (OPS) modulate or eliminate Visual pseudo-Scotomas (VS) induced by auditory stimuli?

Researchers evaluated 38 healthy adults (aged 20-29) using the Vertical Maddox Test to detect functional visual alterations under different conditions. The study included four phases:

* Baseline assessment with no stimuli.
* Assessment with auditory stimuli alone.
* Assessment with simultaneous auditory and Oral Proprioceptive Stimuli (OPS), including tongue/lip positions (Combined Oral Stimuli) and dental pressure/traction stimuli (Dental Stimuli).
* Assessment with Oral Proprioceptive Stimuli (OPS) alone.

Visual pseudo-scotomas were recorded based on participant responses. The study was approved by the local ethics committee and all participants gave informed consent.

DETAILED DESCRIPTION:
Proprioception plays a well-established role in postural control and motor coordination, but increasing evidence supports its involvement in higher-level sensory processing, including spatial localization and multisensory integration. Given the anatomical overlap of trigeminal afferents innervating both oculomotor and orofacial structures, this study focused on the potential interplay between the stomatognathic and visual systems.

This study is an observational investigation with an experimental within-subject design with repeated measures in healthy volunteers.

The aim is to investigate the influence of oral proprioceptive stimuli on visual perception and audiovisual integration in healthy young adults, and explore whether non-invasive oral stimuli could modulate the occurrence of transient visual distortions-specifically Visual pseudo-Scotomas (VS)-when binocular vision is altered, and whether these stimuli could counteract the effects induced by auditory input.

Participants have been screened to ensure normal hearing, vision, and dental status, and underwent testing using the Vertical Maddox Test, which induces a dissociation in binocular vision that relies heavily on proprioceptive cues.

The experimental protocol was composed of four phases:

1. Baseline evaluation with no stimuli.
2. Application of auditory stimuli (500 Hz tones delivered through headphones) to assess their influence on visual perception.
3. Application of simultaneous auditory and Oral Proprioceptive Stimuli (OPS), including both Combined Oral Stimuli (COS, such as specific tongue and lip positions) and Dental Stimuli (DS, consisting of gentle pressure/traction on central incisors using a calibrated probe).
4. Application of Oral Proprioceptive Stimuli (OPS) alone, without sound.

Participants were asked to report the occurrence and location of any Visual pseudo-Scotomas (VS) observed during each phase. These were defined as functional visual field losses detected via the Vertical Maddox Test, with no underlying ocular pathology.

This protocol was developed based on prior work investigating ocular and oral proprioception and its role in multisensory integration. No pharmacological agents, devices, or therapeutic interventions were used. The study is observational in nature, and no biospecimens were collected or retained.

ELIGIBILITY:
EXCLUSION CRITERIA:

* General criteria:

  * Treatment with psychotropic drugs
  * Hearing loss in one or both ears
* Visual criteria:

  * Visual acuity worse than 20/20 in one or both eyes
  * Stereopsis (three-dimensional vision) less than 120 arc sec
  * Vertical phoria greater than 0.75 Δ
  * Strabismus operated on or not
  * Ongoing optometric rehabilitation
  * History of amblyopia
* Dental criteria:

  * Missing one or more incisors
  * Presence of conservative, prosthetic or orthodontic treatment on one or more incisors (fillings, root canal treatments, veneers, crowns, brackets, Invisalign type attachments...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants of the study were healthy young adults recruited among the students of the Faculty of Medicine and Health Sciences of the University of Barcelona, who did not present any of the exclusion criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Presence of Visual Pseudo-Scotomas (VS) under Auditory and/or Oral Proprioceptive Stimulation | During 4-phase experimental protocol (single visit, approx. 45 minutes)
  Participants were assessed for the occurrence of functional visual disturbances (pseudo-scotomas, or VS) during each phase of the protocol using the Vertical Maddox Test. Presence or absence of VS was recorded under three experimental conditions: auditory stimulation alone, combined auditory and oral proprioceptive stimulation, and oral proprioceptive stimulation alone.

SECONDARY OUTCOMES:
Elimination of Sound-Induced Visual Pseudo-Scotomas by Oral Proprioceptive Stimuli | Day 1, during phase 3 (auditory + OPS) of the experimental protocol
  Among participants who experienced VS during auditory stimulation alone, the presence or absence of VS was re-assessed during the combined application of auditory and oral proprioceptive stimuli to determine whether OPS could eliminate sound-induced visual disturbances.
Presence of Visual Pseudo-Scotomas with Oral Proprioceptive Stimulation Alone | Day 1, during phase 4 (OPS alone) of the experimental protocol
  Participants were evaluated for the occurrence of visual pseudo-scotomas under oral proprioceptive stimuli without auditory input, to assess whether OPS alone could induce transient changes in visual perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Odontológico Universitat de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD) that might be shared include anonymized data on age, sex, inclusion/exclusion criteria, and responses related to the presence or absence of visual pseudo-scotomas during each phase of the experimental protocol. Data would be fully de-identified and shared only upon request, under appropriate ethical and legal conditions. At present, no final decision has been made regarding IPD sharing.

REFERENCES:
- [Background] Quercia P, Pozzo T, Marino A, Guillemant AL, Cappe C, Gueugneau N. Alteration in binocular fusion modifies audiovisual integration in children. Clin Ophthalmol. 2019 Jul 4;13:1137-1145. doi: 10.2147/OPTH.S201747. eCollection 2019. PMID 31308621
- [Background] Quercia P, Pozzo T, Marino A, Guillemant AL, Cappe C, Gueugneau N. Children with Dyslexia Have Altered Cross-Modal Processing Linked to Binocular Fusion. A Pilot Study. Clin Ophthalmol. 2020 Feb 13;14:437-448. doi: 10.2147/OPTH.S226690. eCollection 2020. PMID 32103890